CLINICAL TRIAL: NCT06410924
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Evaluate the Efficacy, Safety, and Tolerability of Treatment With DD01 for 48 Weeks in Overweight/Obese Subjects With MASLD/MASH
Brief Title: A Study to Evaluate DD01 in Overweight/Obese Subjects With MASLD/MASH
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Neuraly, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DD01-DN-02
Record Dates: First submitted 2024-05-08; First posted 2024-05-13 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: NAFLD; NASH
Keywords: Liver Disease; Fatty Liver; Non-alcoholic fatty liver disease; Non-alcoholic steatohepatitis; MASH; MASLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Diseases; Fatty Liver

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DD01 (Experimental): Study Drug
  Interventions: Drug: DD01
- Placebo (Placebo Comparator): Matching Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DD01 — Dual GLP-1 and glucagon receptor agonist
  Arms: DD01
Drug: Placebo — Placebo matching DD01
  Arms: Placebo

SUMMARY:
This is a Phase 2 Study to evaluate the effect of DD01 treatment in overweight/obese patients with metabolic dysfunction-associated steatotic liver disease (MASLD)/metabolic dysfunction-associated steatohepatitis (MASH).

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, 18 to 70 years of age
* With MASLD or confirmed diagnosis of MASH based on MRI PDFF ≥10% AND 1 of the following:

  1. Biopsy proven MASH obtained during Screening which confirms the presence of MASH characterized by a NAS ≥4 with at least 1 in each component (steatosis, ballooning, and lobular inflammation) and fibrosis stage F1 to F3. A historical biopsy obtained within 6 months may be acceptable OR
  2. Meets at least 2 additional metabolic syndrome factors
* Participants with a BMI ≥25 kg/m2, with stable body weight by history for 3 months
* Participants must have a waist circumference ≥35 inches (females), or ≥40 inches (males), and must have a waist circumference ≤57 inches (both males and females)
* Female participants must be non-pregnant, non-lactating or post-menopausal
* Participants must have the ability and willingness to comply with all Protocol procedures, provide written informed consent and meet all inclusion criteria as outlined in the study protocol

Exclusion Criteria: Participants who have:

* A history of active or chronic liver disease
* Liver cirrhosis (fibrosis stage F4), any prior history of hepatic decompensation, including low platelet counts, esophageal varices, ascites, hepatic encephalopathy, splenomegaly, any hospitalization for treatment of chronic liver disease, or a Model for End Stage Liver Disease score of ≥12
* Recent (within 3 months of Screening) use of therapies associated with development of MASLD/MASH (eg, systemic corticosteroids, methotrexate, tamoxifen, aromatase inhibitors, amiodarone, or long-term use of tetracyclines)
* Previous surgical treatment for obesity as well as clinically significant GI disorders
* Type 1 diabetes mellitus, or T2DM on insulin and/or GLP-1 receptor agonist therapy, dipeptidyl peptidase-4 inhibitors, or other therapies
* Uncontrolled hypertension or uncontrolled dyslipidemia
* Participated in an investigational study within 30 days prior to dosing or who have participated in another MASLD/MASH interventional study within 60 days prior to Screening
* With a history or current diagnosis of acute or chronic pancreatitis or factors for pancreatitis, symptomatic cholelithiasis and/or choledocholithiasis, or alcohol abuse
* With a history of any major surgery within 3 months prior to Screening
* With heart failure (New York Heart Association Class III or IV) or any cardiovascular event or evidence of active cardiovascular disease
* With a presence of clinically significant 12-lead ECG findings at Screening, or cardiac arrhythmia requiring medical or surgical treatment within 6 months prior to Screening
* With personal or family history of medullary thyroid carcinoma (MTC)
* With a history of renal disease
* With a history of alcohol or illicit drug abuse
* A positive test for hepatitis B surface antigen, hepatitis C RNA, or HIV type 1 or type 2 antibody
* A clinically significant physical examination, ECG, or laboratory finding, as judged by the Investigator, may interfere with any aspect of study conduct or interpretation of results
* Not met any other exclusion criteria as outlined in the study protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2024-06-13 (Actual); Primary Completion 2025-04-22 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects who achieve at least 30% liver fat reduction measured by MRI-PDFF | 12 weeks

SECONDARY OUTCOMES:
Absolute change in percent liver fat content as assessed by MRI-PDFF | 12 weeks and 48 weeks
Change in liver stiffness as assessed by Magnetic Resonance Elastography (MRE) | 12 weeks and 48 weeks
Change in liver stiffness measurements as assessed by FibroScan | 12 weeks and 48 weeks
Change in liver steatosis as assessed by FibroScan | 12 weeks and 48 weeks
Number of participants with Adverse Events | 12 and 48 weeks
Change in liver biochemistry | 12 and 48 weeks
  To determine the effect in liver biochemistry parameters including ALT, AST, AST/ALT ration, Gamma-glutamyl transferase, bilirubin
Change in glucose metabolism parameters | 12 and 48 weeks
  To determine the effect on glucose metabolism parameters including glucose, insulin, C-peptide and HbA1c
Effect on pharmacokinetics as assessed by serum concentration-time profiles | Day 1 to 48 weeks

OTHER OUTCOMES:
Histologic evidence for improvements in MASH | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dennis To, Study Director — Neuraly, Inc.
Locations (11):
- United States (11):
  - Summit Research Site, Maitland, Florida
  - Summit Research Site, Monroe, Louisiana
  - Summit Research Site, West Monroe, Louisiana
  - Summit Research Site, Kansas City, Missouri
  - Summit Research Site, Austin, Texas
  - Summit Research Site, Bellaire, Texas
  - Summit Research Site, Brownsville, Texas
  - Summit Research Site, Corpus Christi, Texas
  - Summit Research Site, Edinburg, Texas
  - Summit Research Site, Georgetown, Texas
  - Summit Research Site, San Antonio, Texas